CLINICAL TRIAL: NCT02844582
Title: A Selective Frontline Cabazitaxel Therapeutic Pathway for Castration-Resistant Prostate Cancer With Integrated Biomarkers
Brief Title: Cabazitaxel and Prednisone in Treating Patients With Metastatic Hormone-Resistant Prostate Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Poor accrual of subjects onto study
Sponsor: University of California, Davis (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 868922; UCDCC#261 (Registry Identifier: UC Davis IRB); UCDCC#261 (Other: University of California Davis Comprehensive Cancer Center); NCI-2016-00961 (Other: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2016-06-28; First posted 2016-07-26 (Estimated); Results first posted 2021-01-25 (Actual); Last update posted 2021-01-25 (Actual); Status verified 2021-01

CONDITIONS: Hormone-Resistant Prostate Cancer; Stage IV Prostate Adenocarcinoma
MeSH Terms: interventions — cabazitaxel; XRP6258; Prednisone; deltacortene; prednylidene

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (cabazitaxel, prednisone) (Experimental): Patients receive cabazitaxel IV over 1 hour on day 1 and prednisone PO BID on days 1-21. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cabazitaxel; Drug: Prednisone

INTERVENTIONS:
Drug: Cabazitaxel — Given IV
  Other Names: Jevtana; RPR-116258A; Taxoid XRP6258; XRP-6258
Drug: Prednisone — Given PO
  Other Names: .delta.1-Cortisone; 1, 2-Dehydrocortisone; Adasone; Cortancyl; Dacortin; DeCortin; Decortisyl; Decorton; Delta 1-Cortisone; Delta-Dome; Deltacortene; Deltacortisone; Deltadehydrocortisone; Deltasone; Deltison; Deltra; Econosone; Lisacort; Meprosona-F; Metacortandracin; Meticorten; Ofisolona; Orasone; Panafcort; Panasol-S; Paracort; PRED; Predicor; Predicorten; Prednicen-M; Prednicort; Prednidib; Prednilonga; Predniment; Prednisonum; Prednitone; Promifen; Servisone; SK-Prednisone

SUMMARY:
This phase II trial studies how well cabazitaxel and prednisone work in treating patients with hormone-resistant prostate cancer that has spread to other parts of the body. Drugs used in chemotherapy, such as cabazitaxel and prednisone, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To test whether men with a poor initial response to androgen deprivation therapy (ADT) have a better front line therapeutic response to cabazitaxel as compared to historical controls of frontline metastatic castrate resistant prostate cancer (CRPC) therapy with abiraterone or enzalutamide.

SECONDARY OBJECTIVES:

I. To determine the Response Evaluation Criteria in Solid Tumors (RECIST) version (v)1.1 response rate, progression free survival (PFS) by Prostate Cancer Clinical Trials Working Group 2 (PCWG2) criteria, and overall survival (OS).

II. To evaluate safety and toxicity profile of cabazitaxel in patients with CRPC.

TERTIARY OBJECTIVES:

I. To collect serum and tumor tissue samples for molecular markers or signature predictive of cabazitaxel benefit (to include status of androgen receptor [AR] pathway, androgen biosynthetic pathway genes, adenosine triphosphate [ATP]-binding cassette sub-family B member 1 [ABCBI], multidrug resistance-associated protein 1 [MRP1], and other mediators of taxane resistance).

OUTLINE:

Patients receive cabazitaxel intravenously (IV) over 1 hour on day 1 and prednisone orally (PO) twice daily (BID) on days 1-21. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed prostate adenocarcinoma
* Metastatic disease
* Able and willing to provide informed consent and to comply with the study procedures
* Castration resistant disease defined as evidence of radiological and/or prostate specific antigen (PSA) progression despite castrate levels of testosterone (serum testosterone < 50 ng/dL [1.7 nmol/L]); for PSA progression, there must be at least 2 sequential rises at a minimum of 1-week intervals; the first PSA value must be >= 4 (Prostate Cancer Working Group 2 [PCWG2] criteria)
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* At least 21 days have passed since completing radiotherapy (exception for radiotherapy: at least 7 days since completing a single fraction of =< 800 cGy to a restricted field or limited-field radiotherapy to non-marrow bearing area such as an extremity or orbit) at the time of registration
* At least 21 days have passed since receiving any investigational agent at the time of registration
* At least 21 days have passed since major surgery
* Neuropathy =< grade 1 at the time of registration
* Has recovered from all therapy-related toxicity to =< grade 2 (except alopecia, anemia and any signs or symptoms of androgen deprivation therapy) at the time of registration
* Poor prognosis disease as defined by any of the following:

  * PSA nadir >=4.0, or
  * Gleason score 8-10, or
  * Time from ADT initiation to CRPC of =< 16 months
* Hemoglobin >= 90 g/L
* Neutrophils >= 1.5 x 10^9 /L
* Platelets >= 100 x 10^9/L
* Aspartate aminotransferase (AST) < 1.5 x upper limit of normal (ULN)
* Alanine aminotransferase (ALT) < 1.5 x ULN
* Bilirubin =< 1.0 x ULN (exceptions for Gilbert's syndrome)
* Creatinine =< 1.5 x ULN

Exclusion Criteria:

* Prior therapy with cabazitaxel or to other drugs formulated with polysorbate 80
* Prior taxanes for CRPC
* Prior enzalutamide, abiraterone or ketoconazole
* Other condition, illness, psychiatric condition, or laboratory abnormality that may increase the risk associated with administration of cabazitaxel, study participation, or may interfere with the interpretation of study results and in the judgment of the investigator would make the patient inappropriate for entry into this study
* Histologic evidence of small cell/neuroendocrine prostate cancer
* Patients with reproductive potential who do not agree to use accepted and effective method of contraception during the study treatment period and up to 6 months after the last administered dose; the definition of "effective method of contraception" will be based on the investigator's judgment

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2017-12-20 (Actual); Primary Completion 2019-06-04 (Actual); Study Completion 2019-06-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Evans, Principal Investigator — University of California, Davis
Locations (1):
- University of California Davis Comprehensive Cancer Center, Sacramento, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Cabazitaxel, Prednisone)
Started | 2
Completed | 2
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Cabazitaxel, Prednisone)
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 2
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: PSA Response Rate, Defined as >= 50% Decline in PSA From Baseline Maintained for at Least 3 Weeks and Measured by the Same Laboratory, and Without Evidence of Other Disease Progression Documented at Time of Confirmatory Values
Description: The response rate will be compared to a historical response rate of 20% using the exact binomial test for a single proportion. Confidence intervals for the response rate will be calculated using Wilson's method.
Time Frame: Up to 18 months.
Population: The study was stopped due to poor accrual, and only 2 patients received study treatment. PSA was collected, but the number of evaluable patients was insufficient to perform analysis of this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Cabazitaxel, Prednisone)
Number analyzed (Participants) | 2
Participants | 0

2. Secondary Outcome: Incidence of Adverse Events, Serious Adverse Events, and Discontinuations, Described and Graded According to the National Cancer Institute Common Terminology Criteria for Adverse Events Version 4.03
Description: Incidence of adverse events, serious adverse events, and discontinuations, described and graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events version 4.03
Time Frame: Up to 28 days after discontinuation of study drug
Measure: Number; unit: participants
Arm/Group | Treatment (Cabazitaxel, Prednisone)
Number analyzed (Participants) | 2
participants
  Back pain | 1
  Diarrhea | 1
  Fatigue | 2
  Hot flashes | 1
  Neutrophil count decreased | 2
  Non-cardiac chest pain | 1
  Pain | 1
  Renal and urinary disorders - Other, specify | 1
  White blood cell decreased | 2

3. Secondary Outcome: Overall Survival (OS) Defined as the Time Interval From the Date of Enrollment to the Date of Death Due to Any Cause.
Description: Confidence intervals for the response rate will be calculated using Wilson's method. Medians will be estimated using the method of Kaplan and Meier, with confidence intervals estimated using Greenwood's method.
Time Frame: Up to 18 months.
Population: Study was terminated prematurely and data was not collected to assess this outcome measure.
Arm/Group | Treatment (Cabazitaxel, Prednisone)
Number analyzed (Participants) | 0

4. Secondary Outcome: Progression-free Survival (PFS) Defined as the Time Interval Between the Date of Enrollment and the Date of the First Documentation by the Prostate Cancer Working Group 2 (PCWG2) Criteria.
Description: as for outcome 3
Time Frame: Approximately 5 months.
Population: Study was terminated prematurely and insufficient data was collected to assess this outcome measure.
Arm/Group | Treatment (Cabazitaxel, Prednisone)
Number analyzed (Participants) | 0

5. Secondary Outcome: Response Evaluation Criteria in Solid Tumors (RECIST) Response Defined as Radiographic Disease Progression
Description: as for outcome 3
Time Frame: Approximately 5 months.
Population: Study was terminated prematurely and insufficient data was collected to assess this outcome measure.
Arm/Group | Treatment (Cabazitaxel, Prednisone)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Up to 28 days after discontinuation of study drug.
Description: Number of Participants with Adverse Events.
Arm/Group | Treatment (Cabazitaxel, Prednisone)
All-Cause Mortality (participants affected / at risk) | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 2/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Cabazitaxel, Prednisone) (N=2)
Back pain (Musculoskeletal and connective tissue disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 2
Headache (Nervous system disorders) | 1
Hot flashes (Vascular disorders) | 1
Neutrophil count decreased (Investigations) | 2
Non-cardiac chest pain (General disorders) | 1
Pain (General disorders) | 1
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 1
White blood cell decreased (Investigations) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-05-23): https://cdn.clinicaltrials.gov/large-docs/82/NCT02844582/Prot_SAP_000.pdf
  • Informed Consent Form (2018-09-10): https://cdn.clinicaltrials.gov/large-docs/82/NCT02844582/ICF_001.pdf